CLINICAL TRIAL: NCT02801227
Title: Oxytocin vs. Prostaglandin for Induction of Labor in Primiparas With Prelabor Rupture of Membrane and Low Bishop Score: Randomized Control Study
Brief Title: Oxytocin vs. Prostaglandin for Induction of Labor in Primiparas With Prelabor Rupture of Membrane and Low Bishop
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Orna Reichman, Dr. Orna Reichman MD MSCE, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0115-16-SZMC
Record Dates: First submitted 2016-06-01; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Premature Rupture of Fetal Membranes
Keywords: premature rupture of membrane; primipara; term; bishop
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Oxytocin; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental)
  Interventions: Drug: Oxytocin
- Prostaglandin E2 (Experimental)
  Interventions: Drug: Prostaglandin E2

INTERVENTIONS:
Drug: Oxytocin — Intravenous oxytocin: 2.5 mIU per minute with increments of 2.5 mIU every 20 minutes until achieving 4-5 contractions during 10 minutes or 20 mIU. Then after continuous infusion without increasing oxytocin dose will be continued. In case of lack of painful contraction/active labor after 24 hours with oxytocin a trial with PGE2 will be initiated (as described for PGE2)
  Arms: Oxytocin
Drug: Prostaglandin E2 — PGE2 2 mg wil be inserted to the posterior fornix, this will be repeated every 6 hours until achieving painful contractions or up to 4 doses (24 hours). In case of lack of painful contraction/active labor after the fourth dose of PGE2 a trial with oxytocin will be initiated (as described for Oxytocin).
  Arms: Prostaglandin E2

SUMMARY:
The purpose of the study is to compare between oxytocin to prostaglandin (PGE2), regarding time from induction of labor (IOL) to delivery among primiparas at term with prelabor rupture of membrane (PROM) and an unfavorable cervix.

DETAILED DESCRIPTION:
The purpose of the study is to compare between oxytocin to prostaglandin (PGE2), regarding time from induction of labor (IOL) to delivery among primiparas at term with prelabor rupture of membrane (PROM) and an unfavorable cervix.

Our secondary outcome is to compare between the groups regarding obstetric complications including: cesarean delivery, operative vaginal delivery, maternal intrapartum fever, postpartum hemorrhage, Apgar score at 5 minutes ≤ 7, PH, admission to NICU and the time from initiation of induction to active labor.

The study population will include primiparous at term with PROM and unfavorable bishop score (≤3). Subsequent to confirming inclusion criteria and after receiving informed consent parturients will be randomly allocated to receive oxytocin or PGE2.

Induction with oxytocin (group 1) will be initiated by infusion of intravenous oxytocin: 2.5 mIU per minute with increments of 2.5 mIU every 20 minutes until achieving 4-5 contractions during 10 minutes. Then after continuous infusion without increasing oxytocin dose will be continued. In case of lack of painful contraction/active labor after 24 hours with oxytocin a trial with PGE2 will be initiated (as described for group 2) Induction with PGE2 (group 2) will be initiated by inserting to the posterior fornix PGE2 2 mg, this will be repeated every 6 hours until achieving painful contractions or up to 4 doses (24 hours). In case of lack of painful contraction/active labor after the fourth dose of PGE2 a trial with oxytocin will be initiated (as described for group1).

Failed induction will be defined for parturients who failed to develop active labor after 48 hours from initiation of induction.

Decisions regarding management of labor including all aspects of labor (augmentation, delivery, postpartum) will be made by the physician in charge and will be based on standards of our labor room.

ELIGIBILITY:
Inclusion Criteria:

Age 18-38 years Primiparas Term (37-42) EFW 2500-4000 PROM < 12 hours Confirmed PROM No painful contractions Vertex presentation Willing to be induced Bishop score: (3 or less) cervix: elongated, posterior, closed, firm-medium, head SP-1 or higher

Exclusion Criteria:

Intrauterine growth retardation preterm<37 weeks painful contraction Other reasons for induction aside from PROM as: severe PIH, uncontrolled GDM Medical conditions that the researcher thinks will affect the outcome

-

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Time from induction of labor to delivery comparing between oxytocin and PGE2 among primiparas with prelabor rupture of membrane at term and low Bishop score (≤ 3) regarding the time needed to complete a vaginal delivery. | up to 48 hours

SECONDARY OUTCOMES:
cesarean delivery | 3 dyas
operative vaginal delivery | 3 dyas
maternal intrapartum fever | one week
postpartum hemorrhage | 3 dyas
Apgar score at 5 minutes ≤ 7 | 3 days
admission to NICU | a week

CONTACTS AND LOCATIONS:
Overall Officials: Orna Reichman, MD, Principal Investigator — Shaare Zedek Medical Center

IPD SHARING:
Plan to Share IPD: Yes